CLINICAL TRIAL: NCT05830838
Title: Daily Adaptive Post-Prostatectomy Radiation With Stereotactic Ablative Radiotherapy (DAPPER)
Brief Title: Daily Adaptive Post-Prostatectomy With Stereotactic Ablative Radiotherapy in Patients With Prostate Cancer
Acronym: DAPPER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Bradley (Brad) Stish, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMROR2251; NCI-2023-02453 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22-006248 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2023-04-01; First posted 2023-04-26 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Malignant Prostate Neoplasm
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (daily adaptive online replanning, SBRT) (Experimental): Patients undergo daily adaptive online replanning for SBRT to the prostate fossa on study. Patients also undergo MRI and may undergo PET/CT during screening.
  Interventions: Procedure: Computed Tomography; Radiation: Image-Guided Adaptive Radiation Therapy; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Radiation: Stereotactic Body Radiation Therapy
- Group II (daily adaptive online replanning, SBRT) (Experimental): Patients undergo daily adaptive online replanning for SBRT to the prostate fossa and pelvic lymph nodes on study. Patients also undergo MRI and may undergo PET/CT during screening.
  Interventions: Procedure: Computed Tomography; Radiation: Image-Guided Adaptive Radiation Therapy; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Radiation: Image-Guided Adaptive Radiation Therapy — Undergo daily adaptive online replanning for SBRT
  Other Names: IGART
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Other: Questionnaire Administration — Ancillary studies
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy

SUMMARY:
This clinical trial evaluates the feasibility, safety, and tolerability of stereotactic ablative radiotherapy (SABR) using daily adaptive radiation techniques to the prostate fossa and/or pelvic lymph nodes in patients with prostate cancer who have undergone surgical removal of the prostate (radical prostatectomy). For patients with prostate cancer who develop a rising prostate specific antigen (PSA) after radical prostatectomy, salvage radiation therapy is the standard of care treatment. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. All patients receiving salvage radiation following radical prostatectomy typically have treatment directed to the prostate fossa, which is the anatomical region around the operative bed that is at highest risk for containing left over tumor. Many patients receiving salvage radiation therapy can also benefit from treatment of the pelvic lymph nodes. Adaptive radiotherapy is an emerging treatment technique that uses daily imaging to adjust treatment volumes, ensure accurate dose delivery, and allow the use of smaller planning target volume margins. Adaptive radiation is ideally suited for the further implementation of SABR treatment regimens directed to the prostate fossa with or without inclusion of the pelvic lymph nodes. While daily adaptive radiation therapy has been reported in other disease settings, there is currently no data about its use for post-prostatectomy radiation. Using daily adaptive radiation techniques may help researchers learn how to minimize exposure to normal tissue and shorten the number of required treatments to better target the radiation dose in prostate cancer patients post-prostatectomy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To demonstrate the safety of daily, adaptive online replanning in patients treated with stereotactic body radiation therapy (SBRT) to the prostate +/- pelvic lymph nodes as defined by observation of a grade 3 genitourinary and gastrointestinal toxicity rate of less than or equal to 5%.

SECONDARY OBJECTIVES:

I. To determine the feasibility of daily, adaptive online replanning for patients receiving SBRT to the prostate fossa +/- pelvic lymph nodes.

II. To assess the efficacy of daily, adaptive SBRT to the prostate fossa. III. To measure the change in patient reported urinary, bowel, and sexual outcomes following protocol treatment.

EXPLORATORY OBJECTIVE:

I. To assess the dosimetric benefits of daily adaptive replanning for prostate fossa/pelvic lymph node SBRT.

OUTLINE: Patients are assigned to 1 of 2 groups.

GROUP I: Patients undergo daily adaptive online replanning for SBRT to the prostate fossa on study. Patients also undergo (MRI) of the prostate fossa and pelvis and may undergo positron emission tomography/computed tomography (PET/CT) during screening.

GROUP II: Patients undergo daily adaptive online replanning for SBRT to the prostate fossa and pelvic lymph nodes on study. Patients also undergo MRI of the prostate fossa and pelvis and may undergo PET/CT during screening.

ELIGIBILITY:
Inclusion Criteria:

* Males age >= 18 years who are receiving post-operative radiation therapy to the prostate fossa, with or without inclusion of the pelvic lymph nodes, for biochemical recurrences after radical prostatectomy.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) =< 2.
* Ability to complete questionnaire(s) by themselves or with assistance.
* Provide written informed consent.
* Willingness and ability to complete protocol-specified follow-up (during the active monitoring phase of the study).

Exclusion Criteria:

* Current evidence of untreated metastatic prostate cancer involving nonregional lymph nodes outside of the bony pelvis, bone, or visceral organs.
* Receipt of cytotoxic chemotherapy within 3 months prior to enrollment.
* Prior radiation therapy to pelvis such that the proposed study treatment volume received 10 Gy or greater.
* Co-morbid severe concurrent disease that would result in a life expectancy of < 5 years.
* Diabetes mellitus-associated vascular ulcers or wounding healing problems, inflammatory bowel disease, or a diagnosed connective tissue disorder.
* Medical or psychiatric conditions that preclude informed decision-making or adherence to study protocols.
* Men of childbearing potential who are unwilling to employ adequate contraception.
* History of a bladder neck contracture, urethral stricture that required dilation, or any surgical repair/reconstruction involving the bladder or urethra other than radical prostatectomy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-07-28 (Actual); Primary Completion 2028-05-30 (Estimated); Study Completion 2029-05-30 (Estimated)

PRIMARY OUTCOMES:
Observe Grade 3 genitourinary and gastrointestinal toxicity rate to demonstrate safety of daily adaptive online replanning | Up to 5 years
  Acute and late Common Terminology Criteria for Adverse Events version 5.0 grade 2 or greater genitourinary and gastrointestinal toxicity will be recorded for all patients. Will report the overall grade 3+ toxicity rate along with a 95% confidence interval for this endpoint. Metrics related to treatment times for each fraction, physician choice of baseline vs adaptive plan, and any potential patient safety issue related to the adaptive planning process will be assessed as well.

SECONDARY OUTCOMES:
Evaluate successful completion of daily adaptive radiation planning | Up to 5 years
  Measured by the successful completion of the daily adaptive radiation planning process, allowing the physician to choose this adaptive plan or the preexisting baseline plan. Successful completion of the daily adaptive radiation planning process will be recorded on a per fraction basis for each patient in the Ethos treatment planning system. Will be met if >= 90% of all fractions are completed. Metrics related to treatment times for each fraction, physician choice of baseline versus (vs) adaptive plan, and any potential patient safety issue related to the adaptive planning process will be assessed as well. Will be reported descriptively, including the overall rates and 95% confidence intervals. The continuous variables will be compared between the groups (baseline vs adaptive plans) using the Wilcoxon Rank-Sum test and categorical variables will associated with the groups via chi-square tests. Graphical methods will be used as well, such as boxplots to display the continuous data
Local failure | From enrollment up to 5 years
  Local failure will be considered to have occurred if the patient develops a biopsy proven or radiographically confirmed site of recurrent disease within a planning target volume at any time following completion of protocol treatment. Patients will be recorded as experiencing an event on the date they were noted to meet the definition for recurrence. Will be reported as cumulative incidence with 95% confidence intervals. All baseline variables will be assessed for correlations with efficacy outcomes using the Wilcoxon Rank-Sum test for continuous variables and chi-square tests for categorical variables. Kaplan-Meier plots will be used as a graphical method to report data.
Biochemical failure | From baseline up to 5 years
  Biochemical failure is defined by prostate specific antigen (PSA) measurements following treatment. A biochemical failure will be declared if a patient's PSA rises more than 0.4 ng/ml above their post-radiation therapy nadir. Biochemical failure can also occur if a patient begins a new prostate cancer-directed therapy following radiation therapy prior to reaching the PSA threshold for biochemical failure. Patients will be recorded as experiencing an event on the date they were noted to meet the definition for recurrence. Will be reported as cumulative incidence with 95% confidence intervals. All baseline variables will be assessed for correlations with efficacy outcomes using the Wilcoxon Rank-Sum test for continuous variables and chi-square tests for categorical variables. Kaplan-Meier plots will be used as a graphical method to report data.
Distant metastasis | From baseline up to 5 years
  Distant metastasis is defined as radiographic or histologic confirmed disease progression within non-regional lymph nodes (M1a), bones, or visceral organs. Patients will be recorded as experiencing an event on the date they were noted to meet the definition for recurrence. Will be reported as cumulative incidence with 95% confidence intervals. All baseline variables will be assessed for correlations with efficacy outcomes using the Wilcoxon Rank-Sum test for continuous variables and chi-square tests for categorical variables. Kaplan-Meier plots will be used as a graphical method to report data.
Assess patient reported changes in urinary, bowel, and sexual outcomes following protocol treatment with the Expanded Prostate Cancer Index Composite-26 (EPIC-26) instrument. | Up to 2 years
  EPIC-26 contains 26 item in 5 domains: Urinary Incontinence, Urinary Irritative/Obstructive, Bowel, Sexual, and Hormonal. Response options for each EPIC item form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale, with higher scores representing better Health Related Quality of Life. Will calculate the number of patients experiencing a minimally important difference (MID). MID will be considered a chance of >0.5 standard deviations from the pre-treatments median score within a specific domain.
Change in patient reported urinary, bowel, and sexual outcomes following protocol treatment with the Expanded Prostate Cancer Index Composite-26 (EPIC-26) instrument. | Baseline, Up to 2 years
  EPIC-26 contains 26 item in 5 domains: Urinary Incontinence, Urinary Irritative/Obstructive, Bowel, Sexual, and Hormonal. Response options for each EPIC item form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale, with higher scores representing better Health Related Quality of Life. Will measure changes in each domain and report these with 95% confidence intervals over time and associate outcomes with baseline variables.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley J. Stish, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials